CLINICAL TRIAL: NCT01108185
Title: Evaluation of the Treatment With Klacid SR in Patients With Acute Tracheitis, Tracheobronchitis and Bronchitis, Acute Exacerbation of Chronic Bronchitis or Mild Community-acquired Bronchopneumonia in Common Clinical Practice in the Slovak Republic
Brief Title: Evaluation of the Treatment With Klacid®SR in Patients With Lower Respiratory Tract Infection
Status: Completed | Type: Observational
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Other Study IDs: P12-060
Record Dates: First submitted 2010-04-20; First posted 2010-04-21 (Estimated); Results first posted 2011-08-25 (Estimated); Last update posted 2011-09-13 (Estimated); Status verified 2011-09

CONDITIONS: Tracheitis; Tracheobronchitis; Bronchitis; Chronic Bronchitis; Community-acquired Pneumonia
Keywords: treatment with Klacid®SR; tracheitis; tracheobronchitis; bronchitis; chronic bronchitis; community-acquired pneumonia
MeSH Terms: conditions — Tracheitis; Bronchitis; Bronchitis, Chronic; Community-Acquired Pneumonia

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Acute Respiratory Infections: Slovak patients with lower respiratory tract infection or patients with acute exacerbation of chronic bronchitis (AECB) or mild community-acquired pneumonia (CAP).

SUMMARY:
The aim of this post-marketing observational study (PMOS) is to describe the relief of symptoms, tolerability and compliance of treatment with Klacid®SR in a dose 1000 mg once daily in patients with lower respiratory tract infection or in patients with acute exacerbation of chronic bronchitis (AECB) or mild community-acquired pneumonia (CAP).

DETAILED DESCRIPTION:
This PMOS will be conducted in a prospective, open-label, single-country, multicenter format. The investigational sites will be consulting rooms of GPs (general practitioner), pneumologists and centers with experience in the treatment of patients with lower respiratory tract infection, AECB (acute exacerbation of chronic bronchitis) and CAP (mild community-acquired pneumonia). Since this will be a PMOS, Klacid®SR will be prescribed in usual manner in accordance with the terms of the local market authorization with regards to dose, population and indication as well as local guidelines. The decision to prescribe or not prescribe Klacid®SR would be taken prior to entry of a subject in the study.

Follow-up of patients should enable two patient visits during this period. Screening/Inclusion Visit will be performed when the decision to start the treatment with Klacid®SR is made. Inclusion of patient in the study will succeed at day 0 (S/I Visit). The Second Visit will follow 10 - 16 days after the Screening/Inclusion Visit.

ELIGIBILITY:
Inclusion Criteria:

* Men, women at least 18 years old

  * with acute tracheitis,
  * acute tracheobronchitis,
  * acute bronchitis,
  * mild community-acquired pneumonia or
  * acute exacerbation of chronic bronchitis

Exclusion Criteria:

* Patients with known hypersensitivity to macrolide antibiotics
* Patients with documented renal impairment (creatinine clearance under 30 ml/min).
* Patients with documented liver parenchyma impairment (AST, ALT and GMT > 3x higher level in comparison with the norm)
* Concomitant therapy with the following drugs: astemizole, cisapride, colchicine, pimozide, terfenadine and ergotamine or dihydroergotamine
* Pregnancy
* Breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients included in this PMOS will be those with acute tracheitis, acute tracheobronchitis, acute bronchitis, mild CAP and acute exacerbation of chronic bronchitis with infectious etiology caused probably by an atypical agent.
Sampling Method: Non-Probability Sample
Enrollment: 3181 (Actual)
Dates: Start 2010-03; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Hloska, M.D., Study Director — Abbott
Locations (158):
- Slovakia (158):
  - Site Reference ID/Investigator# 37753, Banská Bystrica
  - Site Reference ID/Investigator# 37758, Banská Bystrica
  - Site Reference ID/Investigator# 37806, Bardejov
  - Site Reference ID/Investigator# 38052, Bojnice
  - Site Reference ID/Investigator# 37830, Bratislava
  - Site Reference ID/Investigator# 37828, Bratislava
  - Site Reference ID/Investigator# 37823, Bratislava
  - Site Reference ID/Investigator# 37824, Bratislava
  - Site Reference ID/Investigator# 37827, Bratislava
  - Site Reference ID/Investigator# 37826, Bratislava
  - Site Reference ID/Investigator# 37680, Bratislava
  - Site Reference ID/Investigator# 37681, Bratislava
  - Site Reference ID/Investigator# 37825, Bratislava
  - Site Reference ID/Investigator# 37829, Bratislava
  - Site Reference ID/Investigator# 37732, Bratislava
  - Site Reference ID/Investigator# 37831, Bratislava
  - Site Reference ID/Investigator# 37833, Bratislava
  - Site Reference ID/Investigator# 37729, Bratislava
  - Site Reference ID/Investigator# 37840, Bratislava
  - Site Reference ID/Investigator# 37679, Bratislava
  - Site Reference ID/Investigator# 37835, Bratislava
  - Site Reference ID/Investigator# 37839, Bratislava
  - Site Reference ID/Investigator# 37834, Bratislava
  - Site Reference ID/Investigator# 37832, Bratislava
  - Site Reference ID/Investigator# 37678, Bratislava
  - Site Reference ID/Investigator# 37836, Bratislava
  - Site Reference ID/Investigator# 37837, Bratislava
  - Site Reference ID/Investigator# 37838, Bratislava
  - Site Reference ID/Investigator# 37861, Bratislava
  - Site Reference ID/Investigator# 37864, Bratislava
  - Site Reference ID/Investigator# 37866, Bratislava
  - Site Reference ID/Investigator# 25682, Bratislava
  - Site Reference ID/Investigator# 37677, Bratislava
  - Site Reference ID/Investigator# 37754, Brezno
  - Site Reference ID/Investigator# 37755, Brezno
  - Site Reference ID/Investigator# 37756, Brezno
  - Site Reference ID/Investigator# 37863, Dojč
  - Site Reference ID/Investigator# 38048, Dolné Vestenice
  - Site Reference ID/Investigator# 37694, Dolný Kubín
  - Site Reference ID/Investigator# 38029, Drienov
  - Site Reference ID/Investigator# 38056, Dudince
  - Site Reference ID/Investigator# 37688, Galanta
  - Site Reference ID/Investigator# 37703, Galanta
  - Site Reference ID/Investigator# 37808, Giraltovce
  - Site Reference ID/Investigator# 37708, Hôrka nad Váhom
  - Site Reference ID/Investigator# 38054, Hronské Kľačany
  - Site Reference ID/Investigator# 37745, Humenné
  - Site Reference ID/Investigator# 37752, Humenné
  - Site Reference ID/Investigator# 37814, Humenné
  - Site Reference ID/Investigator# 37815, Humenné
  - Site Reference ID/Investigator# 37687, Jelka
  - Site Reference ID/Investigator# 37737, Košice
  - Site Reference ID/Investigator# 37740, Košice
  - Site Reference ID/Investigator# 37741, Košice
  - Site Reference ID/Investigator# 37744, Košice
  - Site Reference ID/Investigator# 37767, Košice
  - Site Reference ID/Investigator# 37788, Košice
  - Site Reference ID/Investigator# 38030, Košice
  - Site Reference ID/Investigator# 38035, Košice
  - Site Reference ID/Investigator# 38040, Košice
  - Site Reference ID/Investigator# 38043, Košice
  - Site Reference ID/Investigator# 37742, Košice
  - Site Reference ID/Investigator# 37810, Levoča
  - Site Reference ID/Investigator# 37811, Levoča
  - Site Reference ID/Investigator# 37686, Likavka
  - Site Reference ID/Investigator# 37790, Lučenec
  - Site Reference ID/Investigator# 37791, Lučenec
  - Site Reference ID/Investigator# 37792, Lučenec
  - Site Reference ID/Investigator# 37793, Lučenec
  - Site Reference ID/Investigator# 37795, Lučenec
  - Site Reference ID/Investigator# 37797, Lučenec
  - Site Reference ID/Investigator# 37798, Lučenec
  - Site Reference ID/Investigator# 37690, Ľubochňa
  - Site Reference ID/Investigator# 37859, Malacky
  - Site Reference ID/Investigator# 37865, Malacky
  - Site Reference ID/Investigator# 37696, Martin
  - Site Reference ID/Investigator# 37702, Martin
  - Site Reference ID/Investigator# 37706, Martin
  - Site Reference ID/Investigator# 37743, Michalovce
  - Site Reference ID/Investigator# 37766, Michalovce
  - Site Reference ID/Investigator# 38028, Michalovce
  - Site Reference ID/Investigator# 37862, Modra
  - Site Reference ID/Investigator# 38042, Moldava nad Bodvou
  - Site Reference ID/Investigator# 37697, Námestovo
  - Site Reference ID/Investigator# 38041, Nitra
  - Site Reference ID/Investigator# 38050, Nitra
  - Site Reference ID/Investigator# 38053, Nitra
  - Site Reference ID/Investigator# 38036, Nitra
  - Site Reference ID/Investigator# 38038, Nitra
  - Site Reference ID/Investigator# 38039, Nitra
  - Site Reference ID/Investigator# 37692, Nitrianske Pravno
  - Site Reference ID/Investigator# 38047, Nitrianske Rudno
  - Site Reference ID/Investigator# 38045, Nováky
  - Site Reference ID/Investigator# 38049, Oslany
  - Site Reference ID/Investigator# 38051, Partizánske
  - Site Reference ID/Investigator# 37731, Piešťany
  - Site Reference ID/Investigator# 37858, Piešťany
  - Site Reference ID/Investigator# 37812, Podhradie
  - Site Reference ID/Investigator# 37757, Pohorelská Maša
  - Site Reference ID/Investigator# 37804, Prešov
  - Site Reference ID/Investigator# 37809, Prešov
  - Site Reference ID/Investigator# 37817, Prešov
  - Site Reference ID/Investigator# 37789, Revúca
  - Site Reference ID/Investigator# 37799, Revúca
  - Site Reference ID/Investigator# 37762, Rimavská Sobota
  - Site Reference ID/Investigator# 37763, Rimavská Sobota
  - Site Reference ID/Investigator# 37764, Rimavská Sobota
  - Site Reference ID/Investigator# 37765, Rimavská Sobota
  - Site Reference ID/Investigator# 37800, Rožňava
  - Site Reference ID/Investigator# 37801, Rožňava
  - Site Reference ID/Investigator# 37698, Ružomberok
  - Site Reference ID/Investigator# 37693, Ružomberok
  - Site Reference ID/Investigator# 37735, Selice
  - Site Reference ID/Investigator# 37733, Senec
  - Site Reference ID/Investigator# 37730, Senica
  - Site Reference ID/Investigator# 38055, Slatina nad Bebravou
  - Site Reference ID/Investigator# 37805, Slovinky
  - Site Reference ID/Investigator# 38033, Snina
  - Site Reference ID/Investigator# 38034, Snina
  - Site Reference ID/Investigator# 38037, Snina
  - Site Reference ID/Investigator# 37746, Spišská Nová Ves
  - Site Reference ID/Investigator# 37747, Spišská Nová Ves
  - Site Reference ID/Investigator# 37748, Spišská Nová Ves
  - Site Reference ID/Investigator# 37750, Spišská Nová Ves
  - Site Reference ID/Investigator# 37751, Spišská Nová Ves
  - Site Reference ID/Investigator# 37813, Spišská Nová Ves
  - Site Reference ID/Investigator# 37736, Streda nad Bodrogom
  - Site Reference ID/Investigator# 38031, Streda nad Bodrogom
  - Site Reference ID/Investigator# 37860, Stupava
  - Site Reference ID/Investigator# 37816, Svidník
  - Site Reference ID/Investigator# 37685, Šamorín
  - Site Reference ID/Investigator# 38046, Topoľčany
  - Site Reference ID/Investigator# 37734, Trenčín
  - Site Reference ID/Investigator# 37699, Trenčín
  - Site Reference ID/Investigator# 37682, Trhová Hradská
  - Site Reference ID/Investigator# 37683, Trhová Hradská
  - Site Reference ID/Investigator# 37691, Trnava
  - Site Reference ID/Investigator# 37705, Trnava
  - Site Reference ID/Investigator# 37870, Trnava
  - Site Reference ID/Investigator# 37701, Trnovec nad Váhom
  - Site Reference ID/Investigator# 37695, Turany
  - Site Reference ID/Investigator# 38032, Veľké Kapušany
  - Site Reference ID/Investigator# 37868, Veľké Kostoľany
  - Site Reference ID/Investigator# 37760, Veľký Krtíš
  - Site Reference ID/Investigator# 37761, Veľký Krtíš
  - Site Reference ID/Investigator# 37807, Vranov nad Topľou
  - Site Reference ID/Investigator# 37867, Vrbové
  - Site Reference ID/Investigator# 37684, Vrútky
  - Site Reference ID/Investigator# 37869, Zohor
  - Site Reference ID/Investigator# 37794, Zvolen
  - Site Reference ID/Investigator# 37796, Zvolen
  - Site Reference ID/Investigator# 37802, Zvolen
  - Site Reference ID/Investigator# 37803, Zvolen
  - Site Reference ID/Investigator# 38044, Žabokreky nad Nitrou
  - Site Reference ID/Investigator# 37689, Žilina
  - Site Reference ID/Investigator# 37700, Žilina
  - Site Reference ID/Investigator# 37704, Žilina
  - Site Reference ID/Investigator# 37707, Žilina

RESULTS

PARTICIPANT FLOW:
Groups:
- Acute Respiratory Infections: Slovak participants with lower respiratory tract infection or patients with acute exacerbation of chronic bronchitis (AECB) or mild community-acquired pneumonia (CAP) prescribed Klacid SR 1000 mg once daily.
Period: Overall Study
Arm/Group | Acute Respiratory Infections
Started | 3181
Per Protocol Population | 3181
Completed | 3154
Not Completed | 27
Not completed — Non-compliance | 15
Not completed — Lost to Follow-up | 12

BASELINE CHARACTERISTICS:
Arm/Group | Acute Respiratory Infections
Number analyzed (Participants) | 3181
Age, Customized [Number; unit: participants]
  Less than 20 years | 50
  20 to 29 years | 411
  30 to 39 years | 873
  40 to 49 years | 787
  50 to 59 years | 538
  60 to 69 years | 331
  70 to 79 years | 130
  80 years or older | 50
  Age not reported | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | NA — Gender not collected in this study
  Male | NA — Gender not collected in this study
Region of Enrollment [Number; unit: participants]
  Slovakia | 3181
Diagnosis [Number; unit: Participants] — The diagnosis of each participant at Baseline.
  Participants
    Acute tracheobronchitis | 926
    Acute bronchitis | 921
    Acute tracheitis | 870
    Acute exacerbation of chronic bronchitis | 281
    Mild community-acquired bronchopneumonia | 183

OUTCOME MEASURES:

1. Primary Outcome: Compliance (Was the Dosage Followed - Yes, no)
Description: Compliance was assessed by asking physicians if participants took their medication as directed and if not, the reason for noncompliance. The number of participants that completed their course of therapy or did not complete due to noncompliance is reported.
Time Frame: Day 10 - 16
Population: The per-protocol population was analyzed.
Measure: Number; unit: Participants
Arm/Group | Acute Respiratory Infections
Number analyzed (Participants) | 3181
Participants
  Completed course of therapy | 3154
  Did not complete (lost to follow-up) | 12
  Did not complete (noncompliance) | 15
  >Participant felt better | 2
  >Diarrhea | 1
  >Reason not reported | 12

2. Primary Outcome: The Tolerability of Klacid SR Will be Assessed by Evaluation of Adverse Events
Description: The number of participants experiencing adverse events, serious adverse events, or adverse events leading to study discontinuation are summarized. See Reported Adverse Events for additional details.
Time Frame: Day 0 through Days 10 - 16
Population: The per-protocol population was analyzed.
Measure: Number; unit: Participants
Arm/Group | Acute Respiratory Infections
Number analyzed (Participants) | 3181
Participants
  Non-serious adverse events (AEs) | 7
  Serious AEs | 0
  Discontinued due to AEs | 0

3. Secondary Outcome: Body Temperature
Description: Body temperature was measured at Day 0 (Baseline) and 10 to 16 days later (Visit 2). Increased body temperature was defined as body temperature greater than or equal to 37 degrees Celsius/98.6 Fahrenheit. The percentage of participants with increased or normal body temperature at Day 0 (Baseline) is summarized.
Time Frame: Day 0
Population: The per-protocol population was analyzed.
Measure: Number; unit: Percentage
Arm/Group | Acute Respiratory Infections
Number analyzed (Participants) | 3181
Percentage
  Body temperature greater than 37 ºC at Day 0 | 84
  Body temperature less than 37 ºC at Day 0 | 15
  Body temperature not reported at Day 0 | 1

4. Secondary Outcome: Body Temperature
Description: Body temperature was measured at Day 0 (Baseline) and 10 to 16 days later (Visit 2). Increased body temperature was defined as body temperature greater than or equal to 37 degrees Celsius/98.6 Fahrenheit. The percentage of participants with increased or normal body temperature at Visit 2 is summarized.
Time Frame: Day 10 - 16
Population: The per-protocol population was analyzed.
Measure: Number; unit: Percentage
Arm/Group | Acute Respiratory Infections
Number analyzed (Participants) | 3181
Percentage
  Body temperature greater than 37 ºC at Visit 2 | 1
  Body temperature less than 37 ºC at Visit 2 | 98
  Body temperature not reported at Visit 2 | 1

5. Secondary Outcome: Cough and Its Character
Description: Participants were evaluated at Day 0 (Baseline) and 10 to 16 days later (Visit 2). The presence of cough and the type of cough (productive or irritating) was determined by the treating physician based on clinical judgment. The number of participants with each type of cough or no cough at Baseline is presented.
Time Frame: Day 0
Population: The per-protocol population was analyzed.
Measure: Number; unit: Participants
Arm/Group | Acute Respiratory Infections
Number analyzed (Participants) | 3181
Participants
  Had irritating cough | 1920
  Had productive cough | 1152
  Did not have cough | 101
  Presence or absence of cough not reported | 8

6. Secondary Outcome: Cough and Its Character
Description: Participants were evaluated at Day 0 (Baseline) and 10 to 16 days later (Visit 2). The presence of cough and the type of cough (productive or irritating) was determined by the treating physician based on clinical judgment. The number of participants with each type of cough or no cough at Visit 2 is presented.
Time Frame: Day 10 - 16
Population: The per-protocol population was analyzed.
Measure: Number; unit: Participants
Arm/Group | Acute Respiratory Infections
Number analyzed (Participants) | 3181
Participants
  Had irritating cough | 164
  Had productive cough | 178
  Did not have cough | 2828
  Presence or absence of cough not reported | 11

7. Secondary Outcome: Dyspnoea
Description: Participants were evaluated at Day 0 (Baseline) and 10 to 16 days later (Visit 2). The treating physicians used their clinical judgment to determine the presence of dyspnoea (difficulty breathing) and whether it occurred while resting or after exertion. The number of participants with each type of dyspnoea or with no dyspnoea at Baseline is presented.
Time Frame: Day 0
Population: The per-protocol population was analyzed.
Measure: Number; unit: Participants
Arm/Group | Acute Respiratory Infections
Number analyzed (Participants) | 3181
Participants
  Had resting dyspnoea | 141
  Had exertional dyspnoea | 634
  Did not have dyspnoea | 2398
  Presence or absence of dyspnoea not reported | 8

8. Secondary Outcome: Dyspnoea
Description: Participants were evaluated at Day 0 (Baseline) and 10 to 16 days later (Visit 2). The treating physicians used their clinical judgment to determine the presence of dyspnoea (difficulty breathing) and whether it occurred while resting or after exertion. The number of participants with each type of dyspnoea or with no dyspnoea at Visit 2 is presented.
Time Frame: Day 10 - 16
Measure: Number; unit: Participants
Arm/Group | Acute Respiratory Infections
Number analyzed (Participants) | 3181
Participants
  Had resting dyspnoea | 12
  Had exertional dyspnoea | 27
  Did not have dyspnoea | 3128
  Presence or absence of dyspnoea not reported | 14

9. Secondary Outcome: Auscultation
Description: Participants were evaluated at Day 0 (Baseline) and 10 to 16 days later (Visit 2). The treating physician used their clinical judgment to determine the presence of abnormal breathing sounds such as wheezing or crackles using auscultation (listening for sounds within the body, usually with a stethoscope in the chest, neck or abdomen). The number of participants with each type of breath sound at Baseline is summarized.
Time Frame: Day 0
Population: The per-protocol population was analyzed.
Measure: Number; unit: Participants
Arm/Group | Acute Respiratory Infections
Number analyzed (Participants) | 3181
Participants
  Normal breath sounds | 917
  Wheezing | 1223
  Crackles | 1030
  Breath sounds not reported | 11

10. Secondary Outcome: Auscultation
Description: Participants were evaluated at Day 0 (Baseline) and 10 to 16 days later (Visit 2). The treating physician used their clinical judgment to determine the presence of abnormal breathing sounds such as wheezing or crackles using auscultation (listening for sounds within the body, usually with a stethoscope in the chest, neck or abdomen). The number of participants with each type of breath sound at Visit 2 is summarized.
Time Frame: Day 10 - 16
Population: The per-protocol population was analyzed.
Measure: Number; unit: Participants
Arm/Group | Acute Respiratory Infections
Number analyzed (Participants) | 3181
Participants
  Normal breath sounds | 3115
  Wheezing | 36
  Crackles | 15
  Breath sounds not reported | 15

ADVERSE EVENTS:
Time Frame: Adverse events were collected through Visit 2 (10 to 16 days).
Description: Adverse events are based on the per-protocol population.
Arm/Group | Acute Respiratory Infections
Serious Adverse Events (participants affected / at risk) | 0/3181
Other Adverse Events (participants affected / at risk) | 7/3181
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acute Respiratory Infections (N=3181)
Diarrhea, abdominal pain (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Vomiting, transient exanthema (Gastrointestinal disorders) | 1 (1)
Headache, nausea, bad taste in mouth (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.